CLINICAL TRIAL: NCT05102591
Title: A Pilot Clinical Trial of a New Neuromodulation Device for Acute Attacks of Migraine in Children and Adolescents Visiting the Emergency Department
Brief Title: A Pilot Clinical Trial of a New Neuromodulation Device for Acute Attacks of Migraine in Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Serena Orr, MD, MSc, FRCPC, Assistant Professor, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: REB21-0408
Record Dates: First submitted 2021-09-28; First posted 2021-11-01 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Migraine Disorders
Keywords: Migraine; Pediatric; Emergency Department; Remote Electrical Neuromodulation
MeSH Terms: conditions — Migraine Disorders; Emergencies | interventions — Ketorolac; Ketorolac Tromethamine; Metoclopramide; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The investigators will carry out a pilot randomized controlled trial (RCT) to determine the feasibility and acceptability of implementing a double-dummy, parallel and crossover RCT protocol. The parallel-group phase was completed from February 22, 2022 to May 15, 2023, and the crossover design phase was completed from May 16, 2023 to March 1, 2024.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, research staff, and clinical staff, including the investigator, research assistant, research nurse, and attending physician, will remain blind to the study interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard-of-Care IV Group (Other): Patients randomised to the standard of care IV group will receive a single, 45-minute stimulation from a sham remote electrical neuromodulation (REN) device, which will not administer the typical electrical stimulation (modulated frequency of ~ 0.083 Hz and a modulated pulse width of 40-550 µs), and will be given a single dose IV ketorolac and IV metoclopramide, at a dose of 0.5 mg/kg (for a maximum 30 mg) and 0.15 mg/kg (for a maximum 10mg), respectively. Metoclopramide will be infused over 15-30 minutes and ketorolac will be administered as a direct IV push over 1-5 minutes.
  Interventions: Drug: Ketorolac; Drug: Metoclopramide; Device: Sham Remote Electrical Neuromodulation Device
- REN Group (Other): Patients randomised to the REN group will receive a single 45-minutes stimulation from the REN device (modulated frequency of 100-120 Hz and a pulse width of 400 µs) and will also receive two doses of normal saline though an IV. Two doses of saline will be used to match the dosage, route of administration, and duration to ketorolac and metoclopramide, as described above in the standard-of-care IV group.
  Interventions: Device: Active Remote Electrical Neuromodulation Device; Drug: Placebo

INTERVENTIONS:
Drug: Ketorolac — Intervention in syringe for target dose of 0.5 mg/kg, maximum 30 mg of ketorolac (1 mL), and administer as a direct IV push over 1-5 minutes
  Other Names: Toradol
  Arms: Standard-of-Care IV Group
Drug: Metoclopramide — Intervention in 50 mL mini bag of normal saline (0.9% NaCl) for target dose of 0.15 mg/kg, maximum 10 mg of metoclopramide (2 mL), and administer as infusion over 15-30 minutes
  Other Names: Maxeran
  Arms: Standard-of-Care IV Group
Device: Active Remote Electrical Neuromodulation Device — The REN device is a battery-powered, wirelessly controlled neuromodulation device that attaches via armband to the upper arm. The REN device is controlled by a smartphone application and administers electrical stimulation to the local C and Aδ nociceptive sensory nerves of the upper arm. This stimulation is achieved using a symmetrical, biphasic, square pulse, modulated at a frequency between 100-120 Hz. Each pulse has a width of 400 µs and the user, via the smartphone application, can adjust the output current to apply a maximum of 40 mA. Each stimulation session occurs over 45 minutes and each device can administer up to 12 stimulation sessions.
  Other Names: Active REN (Nerivio)
  Arms: REN Group
Drug: Placebo — 0.9% NaCl will be administered to participants through IV in identical dosages, methods, and duration as the ketorolac and metoclopramide interventions described above.
  Other Names: Saline
  Arms: REN Group
Device: Sham Remote Electrical Neuromodulation Device — The sham REN device is identical to the active REN device but the stimulation parameters are different, administering a modulated symmetrical biphasic square electrical pulse, modulated frequency of ~0.083 Hz and a modulated pulse width of 40-550 µ. These sham parameters are designed to induce a sensation that will be perceptible to participants, similar to stimulation from the active REN device, but at a frequency that is low enough so as to not modulate the nociceptive sensory nerves.
  Other Names: Sham REN (Sham Nerivio)
  Arms: Standard-of-Care IV Group

SUMMARY:
Migraine is a neurological disease characterized by severe and recurrent headaches. Children and adolescents with migraine often present to the emergency department (ED) with acute attacks, where migraine accounts for up to ~30% of all pediatric ED visits for headache. Based on the limited evidence, many centers have adopted protocols whereby children and adolescents who visit the ED with acute attacks of migraine are treated with an IV neuroleptic (metoclopramide or prochlorperazine) and an IV non-steroidal anti-inflammatory (ketorolac). This combination of interventions is largely considered to be standard of care despite no rigorous evidence to support this practice. Side effect rates with the neuroleptics (metoclopramide or prochlorperazine) are considerable. Therefore, the current standard of care for managing children and adolescents visiting the ED with acute attacks of migraine poses concern to patients and is associated with significant pain and frequent side effects.

Over the past few years, there has been a growth in research investigating the efficacy and safety of non-invasive neuromodulation for the management of acute attacks of migraine. At present, there are several commercially available, non-invasive neuromodulation devices that effectively and safely treat acute attacks of migraine in adults. Because none of these devices have a high level evidence in children, adolescents, nor in the ED setting, there is clinical equipoise as to which device would be most appropriate to study for treating children and adolescents visiting the ED with acute attacks. Throughout our patient engagement work, children and adolescents with migraine have identified that they are interested in trying remote electrical neuromodulation for treating migraine attacks in the ED.

The investigators completed a pilot randomized controlled trial (RCT) to determine the feasibility and acceptability of executing a phase III RCT, in which children and adolescents visiting the ED with acute attacks of migraine were randomized to REN or standard of care IV treatment. The trial had two phases: initially the design was a parallel-group design, and after 14 months of recruitment to that design, an amendment was made to allow participants to cross over to the other treatment arm if the initial intervention was not effective, in a crossover design. This change was made in response to participant and staff feedback around the parallel-group design.

DETAILED DESCRIPTION:
One in ten Canadian children and adolescents suffer from migraine, and visits to the pediatric emergency department (ED) for acute attacks are common, with over 2,500 annual visits in Alberta alone. Evidence-based acute management options for children and adolescents presenting to the ED with acute attacks of migraine are limited. The current standard of care, which comprises a combination of a neuroleptic (metoclopramide) and a non-steroidal anti-inflammatory (ketorolac), has a low level of evidence and is administered through an intravenous (IV) cannula. However, at least half of children and adolescents presenting to the ED with acute attacks of migraine would prefer to avoid an IV, and these standard of care migraine interventions have substantial side effects and costs. The Nerivio remote electrical neuromodulation (REN) device is a novel, non-invasive, wearable REN device that is applied to the arm using an armband and wirelessly controlled by a smartphone software application. REN has established efficacy and safety for the treatment of acute attacks of migraine in adults, and preliminary open-label efficacy and safety data for use in adolescents. Through user engagement efforts, the investigators have identified that children and adolescents with migraine and ED providers are interested in trying REN to treat refractory acute attacks in the ED.

The investigators completed a pilot randomized controlled trial (RCT) that aimed to determine the feasibility and acceptability of implementing a phase III RCT, in which children and adolescents visiting the ED with acute attacks of migraine were randomized to REN, or to standard of care IV treatment in a double-dummy parallel group design phase, followed by a crossover design phase. During the crossover phase, participants were crossed over to the other treatment arm if the initial intervention is not effective. The objectives of the investigators were:

1. To determine the feasibility of comparing REN to the standard of care IV intervention (i.e., a combination of metoclopramide and ketorolac) for the treatment of children and adolescents visiting the ED with acute attacks of migraine.
2. To determine the acceptability of the study design and of using REN to treat children and adolescents visiting the ED with acute attacks of migraine.
3. To gather preliminary efficacy and safety data on the use of REN to treat children and adolescents visiting the ED with acute attacks of migraine (for both the initial assigned intervention and the crossover intervention where applicable).

The investigators employed a pilot RCT to determine the feasibility and acceptability of implementing a double-dummy, parallel and crossover RCT protocol. The controlled trial was completed with two design phases: 1) a parallel-group phase from February 22, 2022 to May 15, 2023, and 2) a crossover design phase from May 16, 2023 to March 1, 2024. The design was switched to a crossover design mid-way through the trial based on feedback from participants and clinical staff around concerns with not being able to receive typical care in a timely manner if randomized to the REN arm in the parallel-group design.

In this pilot study, children and adolescents visiting the ED with acute attacks of migraine were randomized to initially receive either REN or standard of care IV treatment (i.e. a combination of metoclopramide and ketorolac). Each group also received a blinded control (either normal saline through the IV for the REN group, or sham stimulation for the standard of care IV group). Consenting participants were randomized at a 1:1 ratio to either REN or standard of care IV treatment. The allocation sequence was sent to the research pharmacy and was not accessible to anyone involved in the study or patient care. The REN group received active stimulation and normal saline placebo that appeared identical in appearance and volume to the medications given to the comparison group. The comparison group received a combination of pharmaceutical interventions considered to be the standard of care for treating children and adolescents visiting the ED with migraine: IV metoclopramide and IV ketorolac. The comparison group also received sham stimulation that was low enough that it did not induce conditioned pain modulation, the mechanism of action of REN, but it was perceptible and similar to the sensation induced by the REN device. Stimulation for both groups occurred over 45 minutes. In the crossover design phase, participants were assessed 120 minutes following the initial intervention and were crossed over to the other treatment arm if the initial intervention was not effective. Efficacy and safety outcomes were measured at baseline, 60 minutes, and 120 minutes (for both the initial and crossover study interventions as applicable), as well as 48 hours post-intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 8-18 years visiting the Alberta Children's Hospital Emergency Department (ED) with an acute attack of migraine as per criteria B-E of the International Classification of Headache Disorders-3 criteria (ICHD-3):

B. Headache attacks lasting at least 2 hours (untreated or unsuccessfully treated)

C. Headache has at least two of the following four characteristics:

* unilateral location
* pulsating quality
* moderate or severe pain intensity
* aggravation by or causing avoidance of routine physical activity (eg, walking or climbing stairs)

D. Also has least one of the following:

* nausea and/or vomiting
* photophobia and phonophobia

E. Not better accounted for by another diagnosis in the opinion of the treating physician

Criterion A (at least 5 attacks) is not being used in this study because prior research has shown that removing criterion A increases the sensitivity of these criteria in the ED. The patient and their caregiver will also be required to understand spoken and written English. In addition, potential participants will be required to have an upper arm circumference of at least 20 cm to ensure optimal device fit and safety.

Exclusion Criteria:

Exclusion criteria include the following: allergy or contraindication to metoclopramide, ketorolac, or non-steroidal anti-inflammatories; implanted electrical device, congestive heart failure, severe cardiac or cerebrovascular disease, uncontrolled epilepsy (2 or more unprovoked seizures per year), abnormal skin on both upper arms (e.g., cancerous lesion on both upper arms, metallic implants on both upper arms, or abnormal physical sensation in both upper arms), febrile at triage, head trauma in the past 7 days, current secondary headache, previously enrolled in the study, pregnant or lactating.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Serena L Orr, MD, MSc, FRCPC, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Orr SL, Kuziek J, Ali S, Anderson E, Birnie KA, Hershey AD, Khanna P, Kirton A, Sajobi T, Freedman SB. Remote electrical neuromodulation to treat children and adolescents with migraine in the emergency department: A randomized double-dummy pilot trial. Headache. 2025 Jun;65(6):1015-1026. doi: 10.1111/head.14838. Epub 2024 Sep 17. PMID 39290050

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We employed a double-dummy, double-blind, pilot randomized controlled trial initially as a parallel-group design (February 22, 2022 to May 15, 2023), but switched to a crossover design (May 16, 2023 to March 1, 2024) to address participant concerns about not getting typical IV treatment if REN unsuccessful. Receiving the crossover treatment was not required as per protocol. The trial was carried out in a tertiary care pediatric ED at the Alberta Children's Hospital in Calgary, Alberta, Canada.
Pre-assignment Details: During the parallel-group phase, 3 participants provided written informed consent but withdrew prior to being randomized. As such, 22 participants were enrolled in the entire study but 19 of those were randomized to a study treatment. During the crossover phase, participants were not required to receive the crossover treatment if well enough to go home after the initial treatment. Only 2 participants received the crossover treatment (both REN initially and Standard of Care as crossover).
Groups:
- Standard-of-Care IV Group (Parallel Design Phase): Patients recruited during the parallel phase and randomised to the standard of care IV group will receive a single, 45-minute stimulation from a sham remote electrical neuromodulation (REN) device, which will not administer the typical electrical stimulation (modulated frequency of ~ 0.083 Hz and a modulated pulse width of 40-550 µs), and will be given a single dose IV ketorolac and IV metoclopramide, at a dose of 0.5 mg/kg and 0.15 mg/kg, respectively. Metoclopramide will be infused over 15-30 minutes and ketorolac will be administered as a direct IV push over 1-5 minutes.
  Ketorolac: Intervention in syringe for target dose of 0.5 mg/kg, maximum 30 mg of ketorolac (1 mL), and administer as a direct IV push over 1-5 minutes
  Metoclopramide: Intervention in 50 mL mini bag of normal saline (0.9% NaCl) for target dose of 0.15 mg/kg, maximum 10 mg of metoclopramide (2 mL), and administer as infusion over 15-30 minutes
  Sham Remote Electrical Neuromodulation Device: The sham REN device is identical to the active REN device but the stimulation parameters are different, administering a modulated symmetrical biphasic square electrical pulse, modulated frequency of ~0.083 Hz and a modulated pulse width of 40-550 µ. These sham parameters are designed to induce a sensation that will be perceptible to participants, similar to stimulation from the active REN device, but at a frequency that is low enough so as to not modulate the nociceptive sensory nerves.
- REN Group (Parallel Design Phase): Patients recruited during the parallel phase and randomised to the REN group will receive a single 45-minutes stimulation from the REN device (modulated frequency of 100-120 Hz and a pulse width of 400 µs) and will also receive two doses of normal saline though an IV. Two doses of saline will be used to match the dosage, route of administration, and duration to ketorolac and metoclopramide, as described above in the standard-of-care IV group.
  Active Remote Electrical Neuromodulation Device: The REN device is a battery-powered, wirelessly controlled neuromodulation device that attaches via armband to the upper arm. The REN device is controlled by a smartphone application and administers electrical stimulation to the local C and Aδ nociceptive sensory nerves of the upper arm. This stimulation is achieved using a symmetrical, biphasic, square pulse, modulated at a frequency between 100-120 Hz. Each pulse has a width of 400 µs and the user, via the smartphone application, can adjust the output current to apply a maximum of 40 mA. Each stimulation session occurs over 45 minutes and each device can administer up to 12 stimulation sessions.
  Placebo: 0.9% NaCl will be administered to participants through IV in identical dosages, methods, and duration as the ketorolac and metoclopramide interventions described above.
- Standard-of-Care IV Group First, Then REN Group if Applicable (Crossover Design Phase): Patients recruited during the crossover phase and initially randomised to the standard of care IV group during the crossover phase will receive a single, 45-minute stimulation from a sham remote electrical neuromodulation (REN) device, which will not administer the typical electrical stimulation (modulated frequency of ~ 0.083 Hz and a modulated pulse width of 40-550 µs), and will be given a single dose IV ketorolac and IV metoclopramide, at a dose of 0.5 mg/kg (for a maximum 30 mg) and 0.15 mg/kg (for a maximum 10mg), respectively. Metoclopramide will be infused over 15-30 minutes and ketorolac will be administered as a direct IV push over 1-5 minutes.
  At 120-minutes following the initial study intervention, participants will be assessed to see if they feel ready to go home or if they would like to receive the study treatment they did not initially receive(i.e., treatment from the REN Group). This would be a single 45-minutes stimulation from the REN device (modulated frequency of 100-120 Hz and a pulse width of 400 µs) and will also receive two doses of normal saline though an IV. Two doses of saline will be used to match the dosage, route of administration, and duration to ketorolac and metoclopramide, as described above in the standard-of-care IV group.
  The crossover treatment is not required if the participant is considered well enough to go home (as per protocol).
- REN Group First, Then Standard-of-Care IV Group First if Applicable (Crossover Design Phase): Patients recruited during the crossover phase and initially randomised to the REN group during the crossover phase will receive a single 45-minutes stimulation from the REN device (modulated frequency of 100-120 Hz and a pulse width of 400 µs) and will also receive two doses of normal saline though an IV. Two doses of saline will be used to match the dosage, route of administration, and duration to ketorolac and metoclopramide, as described above in the standard-of-care IV group.
  At 120-minutes following the initial study intervention, participants will be assessed to see if they feel ready to go home or if they would like to receive the study treatment they did not initially receive(i.e., treatment from the Standard-of-Care Group). This would be a single, 45-minute stimulation from a sham remote electrical neuromodulation (REN) device, which will not administer the typical electrical stimulation (modulated frequency of ~ 0.083 Hz and a modulated pulse width of 40-550 µs), and will be given a single dose IV ketorolac and IV metoclopramide, at a dose of 0.5 mg/kg (for a maximum 30 mg) and 0.15 mg/kg (for a maximum 10mg), respectively. Metoclopramide will be infused over 15-30 minutes and ketorolac will be administered as a direct IV push over 1-5 minutes.
  The crossover treatment is not required if the participant is considered well enough to go home (as per protocol).
Period: Overall Study
Arm/Group | Standard-of-Care IV Group (Parallel Design Phase) | REN Group (Parallel Design Phase) | Standard-of-Care IV Group First, Then REN Group if Applicable (Crossover Design Phase) | REN Group First, Then Standard-of-Care IV Group First if Applicable (Crossover Design Phase)
Started | 7 | 7 | 3 | 2
Completed | 7 | 7 | 3 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported per arm/group, separately for the parallel phase and crossover phase. No participants received the REN crossover treatment during the crossover phase as they were well enough to go home after the initial IV treatment (as per protocol). Both participants in the "REN Group First" arm of the crossover phase also received the SoC crossover treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard-of-Care IV Group (Parallel Design Phase) | REN Group (Parallel Design Phase) | Standard-of-Care IV Group First, Then REN Group if Applicable (Crossover Design Phase) | REN Group First, Then Standard-of-Care IV Group First if Applicable (Crossover Design Phase) | Total
Number analyzed (Participants) | 7 | 7 | 3 | 2 | 19
Age, Categorical [Count of Participants; unit: Participants] — Age group of participants. Due to the inclusion and exclusion criteria, participants had to be between 8.00 and 18.00 years of age.
  Participants
    <=18 years | 7 | 7 | 3 | 2 | 19
    Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
    >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Reported age of all participants who were enrolled and completed study treatment.
  Standard-of-Care Group: Range = 11 to 17 years REN Group: Range = 13 to 17 years
  years | 13.7 (2.1) | 15 (1.2) | 15.3 (2.1) | 13 (0) | 14.4 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex of participants as recorded by the research nurse.
  Question wording: "Participant sex (what sex was assigned at birth)". Potential responses = Male, Female, Other
  Participants
    Female | 2 | 5 | 2 | 1 | 10
    Male | 5 | 2 | 1 | 1 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race as reported by participants. Question wording: "Are you:". Possible responses: White, South Asian (e.g., East Indian, Pakistani, Sri Lankan), Chinese, Black, Filipino, Arab, Latin American, Southeast Asian (e.g., Vietnamese, Cambodian, Laotian, Thai), West Asian, Korean, Japanese, Other
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 1 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0
    White | 7 | 6 | 2 | 2 | 17
    More than one race | 0 | 0 | 1 | 0 | 1
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Region participants were recruited from. All participants were recruited exclusively in Canada.
  participants
    Canada | 7 | 7 | 3 | 2 | 19
Current attack baseline pain severity [Median (Inter-Quartile Range); unit: units on a scale] — 11-point (0-10) pain numerical rating as reported by the participant.
  Question wording: "On a scale of 0 to 10, what is the level of your pain for this headache?"
  units on a scale | 7 [7 to 8] | 5 [3.5 to 7.5] | 7 [6.5 to 8] | 8 [8 to 8] | 7 [5.5 to 8]
Current attack duration in hours [Median (Inter-Quartile Range); unit: Hours] — Duration of the current migraine attack (converted to "hours") as reported by the participant.
  Questions wording: "How long has the participant had this headache for?"
  Hours | 96 [60 to 240] | 168 [11.5 to 192] | 72 [39.5 to 84] | 168 [120 to 216] | 96 [54 to 216]
Current attack with aura [Count of Participants; unit: Participants] — Number of participants who report having an aura with the current migraine attack.
  Question wording: "Did the participant have any auras (warnings) that today's headache was going to start?"
  Participants | 4 | 1 | 1 | 0 | 6
History of prior attacks with aura [Count of Participants; unit: Participants] — Number of participants who reported having a history of aura with their migraine attacks.
  Question wording: "Does the participant have any auras (warnings) that the headache is going to start?"
  Participants | 5 | 3 | 1 | 0 | 9
Headache frequency in days/month [Median (Inter-Quartile Range); unit: Days per Month] — Frequency of migraine attacks (days per month) as reported by participants.
  Exact question: "How many days per month does the participant have ANY headaches?"
  Days per Month | 6 [5.5 to 10.5] | 7 [3 to 17.5] | 4 [3 to 9.5] | 5 [5 to 5] | 6 [3.5 to 13.5]
Number of participants with continuous headache at baseline [Count of Participants; unit: Participants] — Number of participants who reported having a continuous headache (reported "Daily" or "Always").
  Question wording: "How often do the participant's headaches occur"
  Potential responses: < 1/month, 1-3/month, 1/week, 2-3/week, 4-6/week, Daily, Always, N/A, this is participant's first headache ever, Other
  Participants | 0 | 1 | 0 | 0 | 1
Number of past headache-related ED visits [Number; unit: Counts] — Numbers of headache-related emergency department visits reported by the participant. Only asked to participants who indicate "Yes" to the question "Has the participant been to the emergency department for headache in the past?"
  Question wording: "How many times has the participant been to the emergency department for headache in the past 2 years?"
  Potential responses: 1, 2, 3, 4, 5, 6 or more
  Counts
    None | 3 | 1 | 1 | 0 | 5
    1 | 0 | 0 | 0 | 1 | 1
    2 | 1 | 0 | 0 | 0 | 1
    3 | 0 | 3 | 1 | 1 | 5
    4 | 0 | 1 | 1 | 0 | 2
    5 | 2 | 0 | 0 | 0 | 2
    >=6 | 1 | 2 | 0 | 0 | 3
Took acute intervention at home prior to ED visit [Count of Participants; unit: Participants] — Number of participants who reported taking any acute intervention(s) at home for their current migraine attack.
  Question wording: "What pain medication(s) did you take at home for this headache?"
  Participants | 7 | 7 | 3 | 2 | 19
On a migraine preventive intervention at home [Count of Participants; unit: Participants] — Number of participants who are currently taking any preventive intervention(s) at home.
  Question wording: "What medication(s) or nutraceutical(s) is the participant currently using to PREVENT headaches?"
  Participants | 4 | 4 | 2 | 0 | 10
PedMIDAS Score [Median (Inter-Quartile Range); unit: units on a scale] — Summed score of the Pediatric Migraine Disability Assessment (PedMIDAS) headache disability questionnaire, as completed by participants. The PedMIDAS aims to assess the degree of migraine-related disability in children and adolescents with headache. It is a 6-item scale whereby patients are asked to quantify the number of days of reduced attendance and functioning in the academic, home and extracurricular spheres over the past three months. Minimum score = 0, Maximum score = 240. Larger scores indicate greater migraine-related disability.
  units on a scale | 80 [29 to 126] | 39 [21 to 54] | 61 [45.5 to 62.5] | 49.5 [43.3 to 55.8] | 49 [28 to 63]
Duration of time with headaches in months [Median (Inter-Quartile Range); unit: Months] — How long participants report having any headaches (in months).
  Question wording: "How long has the participant had any type of headache?"
  Months | 48 [36 to 60] | 3 [1.3 to 24] | 72 [60 to 84] | 2.5 [2.3 to 2.8] | 24 [2.5 to 48]

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Recruitment Rate
Description: The primary outcome for this pilot study involves assessment of the feasibility of using the REN device to treat children and adolescents suffering from acute migraine attacks in the ED. The primary feasibility outcome will be determined based on the recruitment rate, defined as the number of participants enrolled per month. Our target is to have an average recruitment rate of 1.5 participants per month. Feasibility will be used as the primary outcome, along with the secondary outcomes, to provide preliminary data to help design and optimize a fully powered, phase III RCT.
  Recruitment rate for both phases of the study are reported to understand if changing to crossover design improved recruitment. We switched to a crossover design strictly to address participant and recruitment concerns around not receiving standard of care migraine treatment if initially randomized to receive REN treatment and such treatment was unsuccessful.
Time Frame: Evaluated monthly and at the end of recruitment (i.e., 2 years or once the final participant has completed the study)
Population: Number of participants who were screened, deemed eligible, and subsequently enrolled. Three (3) participants during the parallel-group design phase withdrew after consent but before being randomized/receiving study treatments. No other participants withdrew during the study.
Measure: Mean (Standard Deviation); unit: participants per month
Groups:
- Parallel-group Design: A parallel-group design was used between February 22, 2022 to May 15, 2023 where participants were randomized to receive either the SoC or REN arm.
- Crossover Design: We switched to a crossover design between May 16, 2023 and March 1, 2024 whereby participants who did not feel well enough to go home 2 hours after study intervention administration was initiated could cross over and receive the interventions of the other group.
Arm/Group | Parallel-group Design | Crossover Design
Number analyzed (Participants) | 17 | 5
participants per month | 1.1 (1.5) | 0.6 (1.0)

2. Secondary Outcome: Reduction in Pain Severity
Description: Reduction in pain severity between baseline and 1-hour, 2 hours, and 48 hours post-interventions. Pain measured on an 11-point Likert scale where 0 = no pain and 10 = worst pain possible, with lower values indicating no/less pain and higher values indicating more pain. Headache pain was only assessed at 48 hours if participants indicated they were currently experiencing a headache and the 48 hours reduction in pain severity outcome does not include participants who crossed over and were exposed to both interventions as we expected them to become unblinded after being exposed to both study treatments; Standard of Care (Initial Treatment) n = 7, REN (Initial Treatment) n = 5.
Time Frame: Difference between baseline and 1 hour, 2 hours, and 48 hours post-intervention.
Population: Treatment data are combined across phases, separated based on treatment given and time given to be consistent with how we specified results would be reported in the protocol (i.e., "...for both the initial assigned intervention and the crossover intervention where applicable"). Participants who received SoC IV at crossover received REN initially, and vice versa. No participants received REN crossover treatment as they were well enough to go home after the initial IV treatment (as per protocol).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Standard-of-Care IV (Initial Treatment; Parallel and Crossover Phases): Patients randomised to initially receive the standard of care IV group will receive a single, 45-minute stimulation from a sham remote electrical neuromodulation (REN) device, which will not administer the typical electrical stimulation (modulated frequency of ~ 0.083 Hz and a modulated pulse width of 40-550 µs), and will be given a single dose IV ketorolac and IV metoclopramide, at a dose of 0.5 mg/kg (for a maximum 30 mg) and 0.15 mg/kg (for a maximum 10mg), respectively. Metoclopramide will be infused over 15-30 minutes and ketorolac will be administered as a direct IV push over 1-5 minutes.
  Ketorolac: Intervention in syringe for target dose of 0.5 mg/kg, maximum 30 mg of ketorolac (1 mL), and administer as a direct IV push over 1-5 minutes
  Metoclopramide: Intervention in 50 mL mini bag of normal saline (0.9% NaCl) for target dose of 0.15 mg/kg, maximum 10 mg of metoclopramide (2 mL), and administer as infusion over 15-30 minutes
  Sham Remote Electrical Neuromodulation Device: The sham REN device is identical to the active REN device but the stimulation parameters are different, administering a modulated symmetrical biphasic square electrical pulse, modulated frequency of ~0.083 Hz and a modulated pulse width of 40-550 µ. These sham parameters are designed to induce a sensation that will be perceptible to participants, similar to stimulation from the active REN device, but at a frequency that is low enough so as to not modulate the nociceptive sensory nerves.
- REN (Initial Treatment; Parallel and Crossover Phases): Patients randomised to initially receive the REN group will receive a single 45-minutes stimulation from the REN device (modulated frequency of 100-120 Hz and a pulse width of 400 µs) and will also receive two doses of normal saline though an IV. Two doses of saline will be used to match the dosage, route of administration, and duration to ketorolac and metoclopramide, as described above in the standard-of-care IV group.
  Active Remote Electrical Neuromodulation Device: The REN device is a battery-powered, wirelessly controlled neuromodulation device that attaches via armband to the upper arm. The REN device is controlled by a smartphone application and administers electrical stimulation to the local C and Aδ nociceptive sensory nerves of the upper arm. This stimulation is achieved using a symmetrical, biphasic, square pulse, modulated at a frequency between 100-120 Hz. Each pulse has a width of 400 µs and the user, via the smartphone application, can adjust the output current to apply a maximum of 40 mA. Each stimulation session occurs over 45 minutes and each device can administer up to 12 stimulation sessions.
  Placebo: 0.9% NaCl will be administered to participants through IV in identical dosages, methods, and duration as the ketorolac and metoclopramide interventions described above.
- Standard-of-Care IV (Crossover Treatment; Crossover Phase): Patients who initially received stimulation from the REN device and two doses of saline, and then crossed over to receive the standard of care IV and a single, 45-minute stimulation from a sham remote electrical neuromodulation (REN) device, which will not administer the typical electrical stimulation (modulated frequency of ~ 0.083 Hz and a modulated pulse width of 40-550 µs), and will be given a single dose IV ketorolac and IV metoclopramide, at a dose of 0.5 mg/kg (for a maximum 30 mg) and 0.15 mg/kg (for a maximum 10mg), respectively. Metoclopramide will be infused over 15-30 minutes and ketorolac will be administered as a direct IV push over 1-5 minutes.
  Participants are assessed 2-hours after the initial study treatment and, if they indicate they are not well enough to go home, would be given the crossover treatment. As such, the crossover treatment was not required.
- REN (Crossover Treatment; Crossover Phase): Patients randomised to initially receive the Standard of Care IV and stimulation from the sham REN device, and then crossed over to receive a single 45-minutes stimulation from the REN device (modulated frequency of 100-120 Hz and a pulse width of 400 µs) and two doses of normal saline through an IV. Two doses of saline will be used to match the dosage, route of administration, and duration to ketorolac and metoclopramide, as described above in the standard-of-care IV group.
  Participants are assessed 2-hours after the initial study treatment and, if they indicate they are not well enough to go home, would be given the crossover treatment. As such, the crossover treatment was not required.
Arm/Group | Standard-of-Care IV (Initial Treatment; Parallel and Crossover Phases) | REN (Initial Treatment; Parallel and Crossover Phases) | Standard-of-Care IV (Crossover Treatment; Crossover Phase) | REN (Crossover Treatment; Crossover Phase)
Number analyzed (Participants) | 10 | 9 | 2 | 0
units on a scale
  1 hour post-intervention | 2.9 (2.9) | 2.1 (1.3) | 3 (0) |
  2 hours post-intervention | 4 (3.5) | 2.4 (1.6) | 3.5 (0.7) |
  48 hours post-intervention: number analyzed (Participants) | 7 | 5 | 0 | 0
  48 hours post-intervention | 3.3 (2.7) | 2.6 (1.5) |  |

3. Secondary Outcome: Number of Eligible Participants Who Are Screened, Enrolled, and Complete All Assessments
Description: This secondary feasibility outcome involves the following: The number of participants who complete all assessments at each time point (baseline, 60, 120 minutes or at discharge if before 120 minutes, and 48-hours; for both the initial assigned intervention and the crossover intervention where applicable).
Time Frame: Evaluated monthly and at the end of recruitment (i.e., 2 years or once the final participant has completed the study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Standard-of-Care IV (Initial Treatment; Parallel and Crossover Phases): Patients randomised to initially receive the standard of care IV group will receive a single, 45-minute stimulation from a sham remote electrical neuromodulation (REN) device, which will not administer the typical electrical stimulation (modulated frequency of ~ 0.083 Hz and a modulated pulse width of 40-550 µs), and will be given a single dose IV ketorolac and IV metoclopramide, at a dose of 0.5 mg/kg (for a maximum 30 mg) and 0.15 mg/kg (for a maximum 10mg), respectively. Metoclopramide will be infused over 15-30 minutes and ketorolac will be administered as a direct IV push over 1-5 minutes.
- Standard-of-Care IV (Crossover Treatment; Crossover Phase): Patients who initially received stimulation from the REN device and two doses of saline, and then crossed over to receive the standard of care IV and a single, 45-minute stimulation from a sham remote electrical neuromodulation (REN) device, which will not administer the typical electrical stimulation (modulated frequency of ~ 0.083 Hz and a modulated pulse width of 40-550 µs), and will be given a single dose IV ketorolac and IV metoclopramide, at a dose of 0.5 mg/kg (for a maximum 30 mg) and 0.15 mg/kg (for a maximum 10mg), respectively. Metoclopramide will be infused over 15-30 minutes and ketorolac will be administered as a direct IV push over 1-5 minutes.
- REN (Crossover Treatment; Crossover Phase): Patients randomised to initially receive the Standard of Care IV and stimulation from the sham REN device, and then crossed over to receive a single 45-minutes stimulation from the REN device (modulated frequency of 100-120 Hz and a pulse width of 400 µs) and two doses of normal saline through an IV. Two doses of saline will be used to match the dosage, route of administration, and duration to ketorolac and metoclopramide, as described above in the standard-of-care IV group.
Arm/Group | Standard-of-Care IV (Initial Treatment; Parallel and Crossover Phases) | REN (Initial Treatment; Parallel and Crossover Phases) | Standard-of-Care IV (Crossover Treatment; Crossover Phase) | REN (Crossover Treatment; Crossover Phase)
Number analyzed (Participants) | 10 | 9 | 2 | 0
Participants | 10 | 9 | 2 |

4. Secondary Outcome: Global Impression of Change
Description: This acceptability outcome involves the following:
  * The proportion of participants who report a global impression of change as "very much improved" or "much improved".
  * Measured on a 7-point Likert scale (Patient Global Impression scale in clinical status; PGI-C) where 1 = "Very much improved", 4 = "No change", and 7 = "Very much worse"
  * Smaller values indicate improvement of overall change while larger values indicate worsening of overall change.
Time Frame: Evaluated for each participant at 2-hours post-intervention, and 48-hours post-intervention
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Standard-of-Care IV (Initial Treatment; Parallel and Crossover Phases) | REN (Initial Treatment; Parallel and Crossover Phases) | Standard-of-Care IV (Crossover Treatment; Crossover Phase) | REN (Crossover Treatment; Crossover Phase)
Number analyzed (Participants) | 10 | 9 | 2 | 0
participants
  2 Hours | 5 | 3 | 1 |
  48 Hours | 5 | 3 | 1 |

5. Secondary Outcome: Study Feedback From Participants and Staff
Description: This acceptability outcome involves the following:
  - Participant feedback regarding study acceptability. Participant feedback measured on 5-point Likert scale (1 = strongly disagree, 5 = strongly agree), where higher values indicate agreement and lower values indicate disagreement. Feedback questions related to study treatments is reported for both treatment groups and combined across treatment groups. Feedback questions related to the research staff and overall study experience is only combined and reported across both groups, rather than being reported for each group separately since these questions don't relate to specific study treatments.
  Feedback from clinical staff was collected after each participant's enrollment but not analyzed as this feedback was free-form and not collected using a scale.
Time Frame: Participant feedback evaluated at 48 hours post-intervention
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Participants: Participants from both SoC and REN treatment groups.
Arm/Group | Standard-of-Care IV (Initial Treatment; Parallel and Crossover Phases) | REN (Initial Treatment; Parallel and Crossover Phases) | Standard-of-Care IV (Crossover Treatment; Crossover Phase) | REN (Crossover Treatment; Crossover Phase) | All Participants
Number analyzed (Participants) | 10 | 9 | 2 | 0 | 19
units on a scale
  I would be interested in using device instead of IV to treat future migraine attacks in the ED. | 3.9 (1) | 3.6 (1) | 3.5 (0.7) |  | 3.7 (1)
  I would be interested in using device with IV to treat future migraine attacks in the ED. | 3.3 (1.1) | 3.3 (1) | 3.5 (0.7) |  | 3.3 (1)
  I would prefer to only use IV to treat future migraine attacks in the ED. | 2.8 (1) | 2.8 (1) | 3 (0) |  | 2.8 (1)
  I would use the device to treat future migraine attacks at home instead of my usual treatment. | 4.2 (0.8) | 3.3 (1.1) | 3 (1.4) |  | 3.8 (1)
  I would use the device to treat future migraine attacks at home with my usual treatment. | 4 (1.1) | 3.7 (0.9) | 3.5 (0.7) |  | 3.8 (1)
  I would only use my usual treatment instead of the device to treat future migraine attacks at home. | 2.5 (0.5) | 2.8 (1.1) | 3 (1.4) |  | 2.6 (0.8)
  If I could, I would bring the device home with me to treat future migraine attacks at home. | 4.4 (0.5) | 3.7 (1) | 4 (0) |  | 4.1 (0.8)
  I understood the study procedures before providing my informed consent to participate.: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18
  I understood the study procedures before providing my informed consent to participate. |  |  |  |  | 4.7 (0.5)
  The research staff took the necessary amount of time to answer all my questions.: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18
  The research staff took the necessary amount of time to answer all my questions. |  |  |  |  | 4.9 (0.3)
  I understood that participation was voluntary.: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18
  I understood that participation was voluntary. |  |  |  |  | 4.9 (0.3)
  I understood that I could withdraw from the study anytime.: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18
  I understood that I could withdraw from the study anytime. |  |  |  |  | 4.7 (0.6)
  I understood the risk(s) involved with participating in the study.: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18
  I understood the risk(s) involved with participating in the study. |  |  |  |  | 4.4 (0.6)
  I understood the possible benefit(s) involved with participating in the study.: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18
  I understood the possible benefit(s) involved with participating in the study. |  |  |  |  | 4.7 (0.5)
  I felt the research staff were approachable when I had questions or concerns.: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18
  I felt the research staff were approachable when I had questions or concerns. |  |  |  |  | 4.8 (0.4)
  I felt the research staff were easy to contact.: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18
  I felt the research staff were easy to contact. |  |  |  |  | 4.6 (0.6)
  I felt the research staff were professional.: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18
  I felt the research staff were professional. |  |  |  |  | 4.7 (0.5)
  I felt the research staff were knowledgeable.: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18
  I felt the research staff were knowledgeable. |  |  |  |  | 4.6 (0.5)
  I felt the research staff were courteous.: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18
  I felt the research staff were courteous. |  |  |  |  | 4.7 (0.5)
  I felt the research staff were sensitive to my needs.: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18
  I felt the research staff were sensitive to my needs. |  |  |  |  | 4.7 (0.5)
  The study went smoothly.: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18
  The study went smoothly. |  |  |  |  | 4.6 (0.6)
  My overall experience was positive.: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18
  My overall experience was positive. |  |  |  |  | 4.6 (0.6)
  I would recommend to others that they consider participation in this study.: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18
  I would recommend to others that they consider participation in this study. |  |  |  |  | 4.7 (0.6)
  If I was aware of another study at the hospital, I would participate if I was eligible and had time.: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18
  If I was aware of another study at the hospital, I would participate if I was eligible and had time. |  |  |  |  | 4.2 (1.1)

6. Secondary Outcome: Number of Participants Reporting Pain Freedom
Description: Number of participants who indicated they were pain free 2-hours post-intervention. Pain measured on an 11-point Likert scale where 0 = no pain and 10 = worst pain possible, with lower values indicating no/less pain and higher values indicating more pain.
Time Frame: 2 hours post-intervention
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard-of-Care IV (Initial Treatment; Parallel and Crossover Phases) | REN (Initial Treatment; Parallel and Crossover Phases) | Standard-of-Care IV (Crossover Treatment; Crossover Phase) | REN (Crossover Treatment; Crossover Phase)
Number analyzed (Participants) | 10 | 9 | 2 | 0
Participants | 4 | 1 | 0 |

7. Secondary Outcome: Number of Participants Reporting Sustained Pain Freedom
Description: Number of participants who indicated they were pain free 2-hours post-intervention and again 48-hours post-intervention. Pain measured on an 11-point Likert scale where 0 = no pain and 10 = worst pain possible, with lower values indicating no/less pain and higher values indicating more pain.
Time Frame: 48 hours post-intervention
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard-of-Care IV (Initial Treatment; Parallel and Crossover Phases) | REN (Initial Treatment; Parallel and Crossover Phases) | Standard-of-Care IV (Crossover Treatment; Crossover Phase) | REN (Crossover Treatment; Crossover Phase)
Number analyzed (Participants) | 10 | 9 | 2 | 0
Participants | 1 | 1 | 0 |

8. Secondary Outcome: Numbers of Participants Reporting a Change in 4-point Pain Severity Scale Between Baseline and 2 Hours Post-intervention
Description: Number of participants who experienced a pain reduction from "severe" or "moderate" severity down to a "mild" or "no pain" severity, or those participants who experienced a pain reduction from "mild" to "no pain" severity between baseline and 2 hours post-intervention. Measured using the 4-point pain severity scale where 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe. Smaller values indicate no/less severe pain and higher values indicate more severe pain.
Time Frame: 2 hours post-intervention
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard-of-Care IV (Initial Treatment; Parallel and Crossover Phases) | REN (Initial Treatment; Parallel and Crossover Phases) | Standard-of-Care IV (Crossover Treatment; Crossover Phase) | REN (Crossover Treatment; Crossover Phase)
Number analyzed (Participants) | 10 | 9 | 2 | 0
Participants | 6 | 5 | 2 |

9. Secondary Outcome: Number of Participants Reporting Sustained Pain Relief
Description: Change from baseline "moderate" to "severe pain" to "mild or "no pain", or change from baseline "mild pain" to "no pain" 2 hours post-intervention, which is sustained to 48 hours post-intervention. Measured using the 4-point pain severity scale where 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe. Smaller values indicate no/less severe pain and higher values indicate more severe pain. Participants who reported they did not have a headache between 2 hours and 48 hours post-intervention were not asked to rate their pain severity and were considered to have no headache pain at 48 hours.
Time Frame: 48 hours post-intervention
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard-of-Care IV (Initial Treatment; Parallel and Crossover Phases) | REN (Initial Treatment; Parallel and Crossover Phases) | Standard-of-Care IV (Crossover Treatment; Crossover Phase) | REN (Crossover Treatment; Crossover Phase)
Number analyzed (Participants) | 10 | 9 | 2 | 0
Participants | 4 | 4 | 1 |

10. Secondary Outcome: Number of Participants Reporting Adverse Events
Description: The number of participants who reported experiencing adverse events and serious adverse events following intervention
Time Frame: Evaluated from time of intervention to 2 hours and 48 hours post-intervention
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard-of-Care IV (Initial Treatment; Parallel and Crossover Phases) | REN (Initial Treatment; Parallel and Crossover Phases) | Standard-of-Care IV (Crossover Treatment; Crossover Phase) | REN (Crossover Treatment; Crossover Phase)
Number analyzed (Participants) | 10 | 9 | 2 | 0
Participants
  2 hours post-intervention | 1 | 0 | 0 | 0
  48 hours post-intervention | 1 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants Reporting Freedom From Most Bothersome Symptom
Description: The number of participants who experienced freedom from their most bothersome symptom (nausea, vomiting, sensitivity to light, or sensitivity to sound).
Time Frame: 2 hours post-intervention
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard-of-Care IV (Initial Treatment; Parallel and Crossover Phases) | REN (Initial Treatment; Parallel and Crossover Phases) | Standard-of-Care IV (Crossover Treatment; Crossover Phase) | REN (Crossover Treatment; Crossover Phase)
Number analyzed (Participants) | 10 | 9 | 2 | 0
Participants | 8 | 3 | 1 |

12. Secondary Outcome: Number of Participants Discharged From the Emergency Department With no Further Intervention
Description: The number of participants discharged from the emergency department with no further intervention other than study intervention
Time Frame: 2 hours post-intervention (after last intervention, following ED discharge)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard-of-Care IV (Initial Treatment; Parallel and Crossover Phases) | REN (Initial Treatment; Parallel and Crossover Phases) | Standard-of-Care IV (Crossover Treatment; Crossover Phase) | REN (Crossover Treatment; Crossover Phase)
Number analyzed (Participants) | 10 | 9 | 2 | 0
Participants | 6 | 4 | 1 |

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and recorded from the start of study treatment administration until completion of the 48-hour follow-up.
Description: Any symptom, sign, illness or experience that develops or worsens in severity during the study, including intercurrent illnesses or injuries. Abnormal results of diagnostic tests are considered if it:
  * results in study withdrawal
  * is associated with a serious adverse event, or with clinical signs or symptoms
  * leads to additional treatment/tests
  * is considered by the PI to be of clinical significance
  No participants received REN as the crossover treatment during the crossover phase.
Groups:
- Standard-of-Care IV (Crossover Treatment; Crossover Phase): Patients who initially received stimulation from the REN device and two doses of saline, and then crossed over to receive the standard of care IV and a single, 45-minute stimulation from a sham remote electrical neuromodulation (REN) device, which will not administer the typical electrical stimulation (modulated frequency of ~ 0.083 Hz and a modulated pulse width of 40-550 µs), and will be given a single dose IV ketorolac and IV metoclopramide, at a dose of 0.5 mg/kg (for a maximum 30 mg) and 0.15 mg/kg (for a maximum 10mg), respectively. Metoclopramide will be infused over 15-30 minutes and ketorolac will be administered as a direct IV push over 1-5 minutes.
  Participants are assessed 2-hours after the initial study treatment and, if they indicate they are not well enough to go home, they are given the crossover treatment. When participants indicate that they feel well enough to go home after initial study treatments, they are not given the crossover treatment.
- REN (Crossover Treatment; Crossover Phase): Patients randomised to initially receive the Standard of Care IV and stimulation from the sham REN device, and then crossed over to receive a single 45-minutes stimulation from the REN device (modulated frequency of 100-120 Hz and a pulse width of 400 µs) and two doses of normal saline through an IV. Two doses of saline will be used to match the dosage, route of administration, and duration to ketorolac and metoclopramide, as described above in the standard-of-care IV group.
  Participants are assessed 2-hours after the initial study treatment and, if they indicate they are not well enough to go home, they are given the crossover treatment. When participants indicate that they feel well enough to go home after initial study treatments, they are not given the crossover treatment. Because all participants randomized to the standard of care IV group for initial treatment felt well enough to go home after initial treatment, no participants received the REN crossover treatment and no participants in this group were at risk for adverse events during this phase of the study.
Arm/Group | Standard-of-Care IV (Initial Treatment; Parallel and Crossover Phases) | REN (Initial Treatment; Parallel and Crossover Phases) | Standard-of-Care IV (Crossover Treatment; Crossover Phase) | REN (Crossover Treatment; Crossover Phase)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 1/10 | 0/9 | 0/2 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard-of-Care IV (Initial Treatment; Parallel and Crossover Phases) (N=10) | REN (Initial Treatment; Parallel and Crossover Phases) (N=9) | Standard-of-Care IV (Crossover Treatment; Crossover Phase) (N=2) | REN (Crossover Treatment; Crossover Phase) (N=0)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Physical/mental restlessness

LIMITATIONS AND CAVEATS:
Our study was conducted during the COVID19 pandemic, the Fall of 2022 "tripledemic", and a shiga-toxin E. Coli outbreak. These events hampered recruitment and our recruitment estimate is likely lower than what we anticipate under 'normal' conditions. Due to delays in the approval process, we had a shorter crossover than the parallel-group phase (9 vs. 15 months). Lastly, 90% of our study participants were White, as such the generalizability of our results is limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT05102591/Prot_SAP_000.pdf